CLINICAL TRIAL: NCT00005962
Title: A Phase II Randomized Trial of Immunologic and Chemotherapeutic Agents for Treatment of Patients With Relapsed or Refractory Acute Myelogenous Leukemia
Brief Title: Comparison of Three Treatment Regimens in Treating Patients With Relapsed or Refractory Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067944; E-4999
Record Dates: First submitted 2000-07-05; First posted 2003-11-05 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — sargramostim; Cyclophosphamide; Cytarabine; Gemtuzumab; Daunorubicin; Topotecan

INTERVENTIONS:
Biological: sargramostim
Drug: cyclophosphamide
Drug: cytarabine
Drug: gemtuzumab ozogamicin
Drug: liposomal daunorubicin citrate
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as gemtuzumab ozogamicin can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining more than one drug or combining monoclonal antibody with chemotherapy may kill more cancer cells. It is not yet known which treatment regimen is more effective for acute myelogenous leukemia.

PURPOSE: Randomized phase II trial to compare the effectiveness of three treatment regimens in treating patients who have relapsed or refractory acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the rates of complete response (CR) and CR without full platelet recovery in patients with relapsed or refractory acute myelogenous leukemia treated with gemtuzumab ozogamicin and cytarabine vs daunorubicin liposomal and cytarabine vs cyclophosphamide, cytarabine, and topotecan.
* Compare the toxicities of these 3 regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by disease status (relapse less than 6 months after first complete response (CR) vs relapse 6-12 months after first CR vs refractory to conventional initial induction chemotherapy (no more than 2 courses) or first reinduction (no more than 1 course) vs second or greater relapse).

* Induction: Patients are randomized to 1 of 3 treatment arms:

  * Arm I: Patients receive cytarabine IV over 2 hours on days 1-4 and gemtuzumab ozogamicin IV over 2 hours on day 5.
  * Arm II: Patients receive daunorubicin liposomal IV over a minimum of 2 hours on days 1-3 and cytarabine IV over 2 hours (beginning immediately after completion of daunorubicin liposomal infusion) on days 1-4.
  * Arm III: Patients receive cyclophosphamide IV over 1 hour every 12 hours on days 1-3, cytarabine IV over 2 hours (beginning immediately after completion of cyclophosphamide infusion) on days 2-6, and topotecan IV continuously on days 2-6.
* Consolidation: Patients who achieve complete remission (CR) receive 1 additional course of induction therapy on the same arm to which they were originally randomized beginning within 4-6 weeks after initial documentation of CR. Patients on arm II receive no additional daunorubicin liposomal if resting ejection fraction is less than 50% preconsolidation. All patients receive sargramostim (GM-CSF) IV over 4 hours or SQ daily beginning 24 hours after completion of consolidation therapy and continuing until blood counts recover.

Patients are followed every 3 months through year 2, every 6 months through year 5, and then annually thereafter until death.

PROJECTED ACCRUAL: A maximum of 150-165 patients (50-55 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven acute myelogenous leukemia of one of the following types:

  * Acute myeloblastic leukemia (FAB type M0, M1, or M2)
  * Acute promyelocytic leukemia (FAB type M3) allowed if ineligible for an ECOG M3 protocol or if no tretinoin or arsenic trioxide therapy is planned
  * Acute myelomonocytic leukemia (FAB type M4)
  * Acute monocytic leukemia (FAB type M5)
  * Acute erythroleukemia (FAB type M6)
  * Acute megakaryocytic leukemia (FAB type M7)
* Must meet 1 of the following criteria:

  * Relapse less than 6 months after first complete remission (CR)
  * Relapse 6-12 months after first CR
  * Refractory to conventional initial induction chemotherapy (no more than 2 courses) or first reinduction (no more than 1 course)

    * Must have marrow documentation of residual leukemia after chemotherapy (for at least 2 weeks duration)
  * Second or greater relapse
* No relapse greater than 1 year after achieving first CR
* Blast cells must be CD33 positive
* Prior CNS leukemia allowed if there is currently documentation of no CNS involvement on CSF examination (i.e., negative CSF by lumbar puncture)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2.0 mg/dL*
* SGOT less than 2 times upper limit of normal* NOTE: *Unless due to leukemia infiltration

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* See Chemotherapy
* No myocardial infarction within the past 3 months
* No significant congestive heart failure
* No significant cardiac arrhythmia
* Cardiac ejection fraction normal by MUGA scan or echocardiogram
* Resting ejection fraction at least 50% or at least 5% increase with exercise
* Shortening fraction at least 24% or normal by echocardiogram

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent organ damage or other medical problems that would precludestudy therapy
* No concurrent evidence (including positive blood or deep tissue cultures or stains) of invasive fungal infection
* No hypersensitivity to ingredients of gemtuzumab ozogamicin or daunorubicin liposomal
* No other active tumor that would interfere with study therapy or increase risk

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior gemtuzumab ozogamicin

Chemotherapy:

* See Disease Characteristics
* See Biologic therapy
* No prior daunorubicin liposomal or topotecan
* Prior doxorubicin (no greater than 300 mg/m2), daunorubicin (no greater than 300 mg/m2), idarubicin (no greater than 100 mg/m2), or mitoxantrone (no greater than 100 mg/m2) allowed if left ventricular function is adequate
* At least 4 weeks since prior chemotherapy except patients who are refractory to conventional initial induction chemotherapy
* Prior hydroxyurea allowed within 4 weeks prior to beginning study
* Hydroxyurea must be discontinued at least 24 hours prior to beginning study

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy except patients who are refractory to conventional initial induction chemotherapy

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10-04 (Actual); Primary Completion 2005-10 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Litzow, MD, Study Chair — Mayo Clinic
Locations (65):
- United States (62):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Result] Litzow MR, Othus M, Cripe LD, Gore SD, Lazarus HM, Lee SJ, Bennett JM, Paietta EM, Dewald GW, Rowe JM, Tallman MS; Eastern Cooperative Oncology Group Leukemia Committee. Failure of three novel regimens to improve outcome for patients with relapsed or refractory acute myeloid leukaemia: a report from the Eastern Cooperative Oncology Group. Br J Haematol. 2010 Jan;148(2):217-25. doi: 10.1111/j.1365-2141.2009.07917.x. Epub 2009 Oct 5. PMID 19804455
- [Result] Litzow MR, Goloubeva O, Rowe J, et al.: A randomized phase II trial of gemtuzumab ozogamicin vs. liposomal daunorubicin vs. cyclophosphamide plus topotecan, each combined with intermediate dose Ara-C for the treatment of patients with relapsed or refractory acute myelogenous leukemia . [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2359, 2003.